CLINICAL TRIAL: NCT02343757
Title: Alzheimer's Disease Imaging With PET/MRI - Beta-amyloid
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough patient enrollment
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 12-12-13
Record Dates: First submitted 2014-05-08; First posted 2015-01-22 (Estimated); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Dementia; Alzheimer Disease
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PET/CT vs. PET/MRI (Other): Patients will be included if presenting with the clinical suspicious of AD, Mild Cognitive Impairment (MCI) or other cognitive impairment to be further determined.
  Patients will undergo two doubles scans in two steps with a maximum of 2 week between both: the first step will be one day double scan with FDG imaged by PET-CT and PET-MRI; and the second step will be one day double scan with 18F-florbetapir imaged by PET-CT and PET-MRI at a different timepoints as shown in figure 1.
  Interventions: Device: PET/MRI

INTERVENTIONS:
Device: PET/MRI

SUMMARY:
The early detection of a preclinical AD or early stage of AD with amyloid imaging could improve the diagnosis and provide knowledge for better therapeutical approach by combining the best of imaging: structural MR sequences and newly FDA-approved biomarker for amyloid PET imaging, all these two techniques with their strengths in one machine.

Specific Aims and Hypotheses can be summarized as follows:

1. To assess image quality and diagnostic performance of 18F-florbetapir (AMYVID) PET/MRI, including direct comparison to corresponding PET/CT images of the same patients.
2. To evaluate the incremental value of using 18F-florbetapir (AMYVID) in addition to 2-[F-18]-fluoro-2 deoxy-D-glucose (FDG) versus FDG alone. Does quantification of plaque burden correlate with degree of neuronal degeneration as depicted by FDG as well as with clinical severity?
3. To determine plaque burden quantitatively with 18F-florbetapir (AMYVID) in PET (form PET/CT and from PET/MR) using novel software developed specifically for these brain application; Computer-Aid Diagnosis for Dementia for amyloid imaging - CAD4D-amyloid

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected AD, MCI and other cognitive impairment will be referred by their neurologist to have a clinical ordered FDG-PET/CT and clinically indicated AMYVID in addition,
* Patients equal to or greater than 21 years old,
* Signed informed consent by patient or legal guardian,
* Physically capable to cooperate.

Exclusion Criteria:

* Subjects who do not meet the above mentioned inclusion criteria,
* Subjects unwilling or unable to sign the informed consent form,
* Subjects with any significant psychiatric or neurologic disorder or disease other than dementia expected to interfere with the study,
* Subjects unable to undergo MR scanning due to exclusion via UHCMC MR restrictions (e.g. certain implanted metallic or electronic devices),
* History of adverse events related to a previous MR or PET/CT,
* Pregnant women,
* Minors.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2016-11-09 (Actual); Study Completion 2016-11-09 (Actual)

PRIMARY OUTCOMES:
To assess image quality and diagnostic performance of 18F-florbetapir (AMYVID) PET/MRI, including direct comparison to corresponding PET/CT images of the same patients. | within one year
  To assess image quality and diagnostic performance of 18F-florbetapir (AMYVID) PET/MRI, including direct comparison to corresponding PET/CT images of the same patients.

SECONDARY OUTCOMES:
To evaluate the incremental value of using 18F-florbetapir (AMYVID) in addition to 2-[F-18]-fluoro-2 deoxy-D-glucose (FDG) versus FDG alone. | within one year
  2. To evaluate the incremental value of using 18F-florbetapir (AMYVID) in addition to 2-[F-18]-fluoro-2 deoxy-D-glucose (FDG) versus FDG alone. Does quantification of plaque burden correlate with degree of neuronal degeneration as depicted by FDG as well as with clinical severity?
To determine plaque burden quantitatively with 18F-florbetapir (AMYVID) in PET (form PET/CT and from PET/MR) using novel software developed specifically for these brain application; | within one year
  3. To determine plaque burden quantitatively with 18F-florbetapir (AMYVID) in PET (form PET/CT and from PET/MR) using novel software developed specifically for these brain application; Computer-Aid Diagnosis for Dementia for amyloid imaging - CAD4D-amyloid (Philips Research, Hamburg)

OTHER OUTCOMES:
Measurement of Effect (ability of 18F-florbetapir (AMYVID) PET/MRI to assess the diagnosis of a patient, compared to both PET/CT and the diagnosis from the clinical record) | within one year
  The main effect that will be evaluated in this study is the ability of 18F-florbetapir (AMYVID) PET/MRI to assess the diagnosis of a patient, compared to both PET/CT and the diagnosis from the clinical record. Another effect that will be evaluated is if there is an added value when using 18F-florbetapir (AMYVID) in addition to 2-[F-18]-fluoro-2 deoxy-D-glucose (FDG) versus using only FDG in the evaluation of cognitive impairment patients.

CONTACTS AND LOCATIONS:
Overall Officials: James K O'Donnell, MD, Principal Investigator — Unviversity Hospitals Case Medical Center
Locations (1):
- University Hospital Case Medical Center, Cleveland, Ohio, United States